CLINICAL TRIAL: NCT01644695
Title: Repair of Complex Recurrent Incisional Hernias With The Bony Anchoring Reinforcement System (BARS)
Brief Title: Review of Complex Recurrent Hernia Repair
Acronym: BARS
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Institute For Advanced Reconstruction (Other)
Responsible Party: Sponsor
Other Study IDs: BARS
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Results first posted 2012-10-15 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-09

CONDITIONS: Recurrent Hernia
Keywords: BARS; Bony Anchoring Reinforcement System; Hernia; Incisional; Recurrent; abdominal wall reconstruction; abdominal wall defect; mesh; component separation
MeSH Terms: conditions — Hernia; Surgical Wound; Recurrence | interventions — Polypropylenes; AlloMax; Alloderm; strattice; Permacol

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Candidate for BARS procedure.: The subjects selected for this trial were over 18 years of age with an appropriate complex, incisional hernia. These patients were consented and treated with the BARS(bony anchoring reinforcement system)procedure.
  Interventions: Procedure: Bony Anchoring Reinforcement System

INTERVENTIONS:
Procedure: Bony Anchoring Reinforcement System — Abdominal exposure was obtained via a lower horizontal incision, a vertical incision, or through a combination horizontal/vertical (ie fleur-di-lis) pattern. Exploratory laparotomy, lysis of intra-abdominal adhesions with hernia sac excision was performed prior to fascial closure. Primary closure of the abdominal fascia was performed with a combination of components separation and placement of biologic mesh over the fascial incision line in onlay fashion. Typically three bone anchors were used to secure the synthetic mesh at the pubic symphysis and two bone anchors to the ASIS bilaterally. The superior aspect of the marlex mesh was sutured to fascia avoiding any incorporation of the costal perichondrium. Quilting sutures were used to secure the mesh to the rest of the abdominal fascia.
  Other Names: Mytec; Fasten; Marlex; Allomax; Alloderm; Strattice; Permacol

SUMMARY:
Abdominal wall incisional hernia is a common finding in patients who have undergone previous intra-abdominal surgeries. Common methods of abdominal fascial closure include primary closure, mesh inlay versus onlay, with or without component separation. All these methods have been shown to have recurrence rates for hernia between 3%-60% in the literature. The study describes the investigators innovative and preferred method for reconstruction of the abdominal wall as BARS (bony anchoring reinforcement system). This method manages the abdominal fascial integrity to reduce the recurrence of incisional hernia while providing an aesthetically superior abdominal wall contour.

DETAILED DESCRIPTION:
• Overview of Research

* 100 anticipated subjects
* Data collection methods- Patients will be evaluated with serial history and physical exams, as well as EMG evaluations. Patients will be asked to report their degree of function and satisfaction.
* Data analysis methods -Data that we will collect from patients will serve as anecdotal evidence to support the research theory.
* We will collect data from patients from testings conducted at the hospital and private office. We will be conducting pre-testing, post-testing, compare results, and surveys.
* The anticipated significance of this research study is that this procedure may greatly improve the quality of life of these severely debilitated patients, reduce the morbidity and mortality rates, and reduce the health care cost burden of chronic care and recurrent hospitalizations.
* The BARS technique for incisional hernia reconstruction provides excellent reinforcement with improved contour, decreased recurrence rates and decreased morbidity for the abdominal wall.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with recurrent abdominal wall incisional hernias
2. Age > 18
3. No medical contraindications to immunosuppressive therapy (in cases utilizing allograft)
4. Ability and motivation to follow up appropriately
5. Ability and motivation to adhere to rehabilitation regimen
6. Stable sequelae of initial CNS insult

Exclusion Criteria: Minors

1. Pregnancy
2. Major medical or psychiatric illness, which in the investigator's opinion would prevent completion of treatment and interfere with follow-up.
3. Patient unable to tolerate surgery, rehabilitation, or immunosuppressive therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Over 18 with Hernia. Included men and women, minorities, and non-english speakers.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2011-10; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew I Elkwood, MD, Principal Investigator — Institute For Advanced Reconstruction
Locations (1):
- Institute For Advanced Reconstruction, Shrewsbury, New Jersey, United States

REFERENCES:
- [Background] Tong WM, Hope W, Overby DW, Hultman CS. Comparison of outcome after mesh-only repair, laparoscopic component separation, and open component separation. Ann Plast Surg. 2011 May;66(5):551-6. doi: 10.1097/SAP.0b013e31820b3c91. PMID 21346524
- [Background] Ramirez OM, Ruas E, Dellon AL. "Components separation" method for closure of abdominal-wall defects: an anatomic and clinical study. Plast Reconstr Surg. 1990 Sep;86(3):519-26. doi: 10.1097/00006534-199009000-00023. PMID 2143588
- [Background] Hawn MT, Snyder CW, Graham LA, Gray SH, Finan KR, Vick CC. Long-term follow-up of technical outcomes for incisional hernia repair. J Am Coll Surg. 2010 May;210(5):648-55, 655-7. doi: 10.1016/j.jamcollsurg.2009.12.038. PMID 20421023
- [Background] Bisgaard T, Kehlet H, Bay-Nielsen MB, Iversen MG, Wara P, Rosenberg J, Friis-Andersen HF, Jorgensen LN. Nationwide study of early outcomes after incisional hernia repair. Br J Surg. 2009 Dec;96(12):1452-7. doi: 10.1002/bjs.6728. PMID 19918863
- [Background] Sisco M, Dumanian GA. A simple technique to anchor prosthetic mesh to bone. Plast Reconstr Surg. 2005 Dec;116(7):2059-60. doi: 10.1097/01.prs.0000192622.53848.3a. No abstract available. PMID 16327650
- [Background] Francis KR, Hoffman LA, Cornell C, Cortese A. The use of Mitek anchors to secure mesh in abdominal wall reconstruction. Plast Reconstr Surg. 1994 Feb;93(2):419-21. doi: 10.1097/00006534-199402000-00034. PMID 8310039

RESULTS

PARTICIPANT FLOW:
Groups:
- Candidate for BARS Procedure.: The subjects selected for this trial were over 18 years of age with an appropriate complex, incisional hernia. These patients were consented and treated with the BARS(bony anchoring reinforcement system)procedure.
  Bony Anchoring Reinforcement System : Abdominal exposure was obtained via a lower horizontal incision, a vertical incision, or through a combination horizontal/vertical (ie fleur-di-lis) pattern. Exploratory laparotomy, lysis of intra-abdominal adhesions with hernia sac excision was performed prior to fascial closure. Primary closure of the abdominal fascia was performed with a combination of components separation and placement of biologic mesh over the fascial incision line in onlay fashion. Typically three bone anchors were used to secure the synthetic mesh at the pubic symphysis and two bone anchors to the ASIS bilaterally. The superior aspect of the marlex mesh was sutured to fascia avoiding any incorporation of the costal perichondrium. Quilting sutures were used to
Period: Overall Study
Arm/Group | Candidate for BARS Procedure.
Started | 85
Completed | 85
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Candidate for BARS Procedure.
Number analyzed (Participants) | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 85
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 53.25 (10.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 85

OUTCOME MEASURES:

1. Primary Outcome: Recurrence Rate
Description: Evidence of complex incisional hernia recurrence after treatment with BARS procedure.
Time Frame: ongoing, average 2.4 years
Population: Subjects were chosen per protocol according to their candidacy for the BARS procedure. All patients were monitored closely following the operation.
Measure: Number; unit: participants
Arm/Group | Candidate for BARS Procedure.
Number analyzed (Participants) | 85
participants | 3

2. Secondary Outcome: Intra and Post-Operative Complications
Description: Record of intra and post operative complications resulting from BARS(bony anchoring reinforcement system) procedure including but not limited to scarring, pain, numbness, intra-abdominal injury, bleeding, death, infection, anesthesia complications, and need for further surgery.
Time Frame: ongoing, average 2.4 years
Population: There were 6 instances of wound dehiscence. There were 2 instances each of infection, necrosis, DVT,hematoma, and neuroma. There was 1 instance each of cellulitis, bowel obstruction, entrapped nerve, and temporary numbness. Further surgery was required 7 times, of which 3 included partial removal of the mesh. 27 complications in total.
Measure: Number; unit: participants
Arm/Group | Candidate for BARS Procedure.
Number analyzed (Participants) | 85
participants | 27

ADVERSE EVENTS:
Time Frame: Adverse event data was collected with regular, ongoing follow up visits. Average time was 2.4 years.
Groups:
- All Participants: No participant was excempt from this measure.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/85
Other Adverse Events (participants affected / at risk) | 27/85
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=85)
Wound Dehiscence (Skin and subcutaneous tissue disorders) | 6 (6)
Infection (Infections and infestations) | 2 (2)
Necrosis (Musculoskeletal and connective tissue disorders) | 2 (2) — Around injury site.
Hematoma (Skin and subcutaneous tissue disorders) | 2 (2)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
DVT (Blood and lymphatic system disorders) | 2 (2)
Bowel obstruction (Gastrointestinal disorders) | 1 (1)
Neuroma (Nervous system disorders) | 2 (2)
Infected Mesh (Injury, poisoning and procedural complications) | 3 (3)
Drain Issue (Injury, poisoning and procedural complications) | 2 (2)
Entrapped Nerve (Nervous system disorders) | 1 (1)
Neuralgia Paresthetica (Nervous system disorders) | 1 (1)
Further Surgery Required (Injury, poisoning and procedural complications) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No